CLINICAL TRIAL: NCT01450592
Title: Epidemiological Study to Evaluate the Dietary Composition of Indian Type-2 Diabetic Patients Compared to Non-diabetic Population
Brief Title: Study To Assess the Dietary Carbohydrate Content of Indian Diabetic Population
Acronym: STARCH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15922; NN1120IN (Other: Company Internal)
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Last update posted 2013-12-30 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Disease; Diabetes Mellitus
Keywords: Carbohydrate, Dietary
MeSH Terms: conditions — Metabolic Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1
  Interventions: Other: No drug
- Group 2
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — Diabetic Population
  Groups: Group 1
Other: No drug — Non-Diabetic Population
  Groups: Group 2

SUMMARY:
The study is designed as an interventional (as blood investigations will be done) dietary survey of diabetic & non-diabetic population sample of India to understand & compare dietary patterns among them.The study objective is to find out amount of carbohydrate content of daily diet of diabetic population study . This study does not intend to study the effect of any drugs. There will be 2 groups : Type 2 diabetics and non diabetic population. The study will begin after the study approval by ethics committee. The subject will involved after they sign the consent form. The study involves general examination of patients, collection of data like history of disease, interview by dietitian with the help of questionnaire, blood investigations (only in diabetic population only) and glycaemic control status of only diabetic population.The study is planned to be enroll 800 subjects (400 in each groups) from 10 study centers spread across India. The study data will be analyzed with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Population
* Patients willing to provide signed & dated informed consent and comply with study
* Indian diabetic population diagnosed with T2DM for at least 12 months
* Male and non pregnant female with age18 years or more

  * Non-Diabetic Population
* Indian non-diabetic population who are not following any diet plan or dietary advice
* Patients willing to provide signed & dated informed consent and comply with study requirements.
* Male and non pregnant female with age 18 years or more
* Non-diabetic population should be matched in terms of age, sex and centre

Exclusion Criteria:

* Patient unwilling to comply with the study procedures.
* Pregnant & lactating women
* History of cardiovascular event within the previous six months.
* Patients with specific co morbidities, which may impact the patients diet, e.g malignant diseases, advanced dementia, Parkinson's disease and others.
* Suffering from chronic diseases including but not limited to chronic renal failure, chronic liver disease that might interfere with participation in the study as per physician discretion.
* Patients on weight management plan e.g. low carbohydrate diet which includes dietary modifications or dietary alterations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type-2 diabetic and non-diabetic population
Sampling Method: Probability Sample
Enrollment: 796 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percentage of total energy intake as carbohydrate by Indian diabetic population | 1 day
Percentage of complex carbohydrate intake from total carbohydrate by Indian diabetic population | 1 day

SECONDARY OUTCOMES:
Difference in the percentage of total energy intake as carbohydrate by diabetic versus non-diabetic population | 1 day
Difference in the percentage of complex carbohydrate content of diabetic versus non-diabetic population | 1 day
Difference in the percentage of total energy intake as proteins & fats by diabetics versus non-diabetic population | 1 day
Percentage of diabetics population who follows diet plan | 1 day
Percentage of diabetic population with glycaemic control | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, India

REFERENCES:
- [Derived] Joshi SR, Bhansali A, Bajaj S, Banzal SS, Dharmalingam M, Gupta S, Mukhopadhyay S, Shah PR, Sahay R, Sarkar S, Manjrekar PV, Rathod RT, Joshi SS. Results from a dietary survey in an Indian T2DM population: a STARCH study. BMJ Open. 2014 Oct 31;4(10):e005138. doi: 10.1136/bmjopen-2014-005138. PMID 25361834